CLINICAL TRIAL: NCT01958151
Title: Does Pre-procedural Anxiety Affect the Consumption of Sedatives During Colonoscopy?
Brief Title: Pre-procedural Anxiety and Sedation.
Status: Completed | Type: Observational
Sponsor: Basak Ceyda MECO (Other)
Responsible Party: Sponsor-Investigator, Basak Ceyda MECO, MD,DESA, Ankara University
Organization: Ankara University (Other)
Other Study IDs: 10-306-12
Record Dates: First submitted 2013-09-25; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Anxiety
Keywords: colonoscopy; deep sedation; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sedated colonoscopy: Planned colonoscopies for screening under propofol sedation titrated to reach a bispectal index value of 60.
  Anxiety levels are assessed before the procedure with State-Trait Anxiety Inventory Scores.
  Interventions: Other: State-Trait Anxiety Inventory Scores

INTERVENTIONS:
Other: State-Trait Anxiety Inventory Scores — Patients are evaluated before the procedure with State-Trait Anxiety Inventory scores to determine the anxiety level.

SUMMARY:
Colonoscopy is an outpatient procedure performed frequently as a screening test for diagnosis and treatment of a wide range of gastrointestinal problems. It is often viewed as an invasive procedure with the potential for embarrassment, discomfort, and worry. Such fears can result in anxiety that may decrease the tolerance and cooperation of the patient, limit the success of the procedure, and increase the likelihood of complications. Therefore, colonoscopy is frequently performed under sedation. The anxiety level of the patient before the procedure may increase the requirement for sedation. It is important for the anesthesiologist to predict the effective dosages of sedation before the procedure to ensure rapid and comfortable sedation as well as prompt recovery and discharge of the patient.

This prospective cohort study is planned to evaluate the effects of pre-procedural anxiety level on the dose of propofol needed for patient and surgeon satisfaction during colonoscopy.

DETAILED DESCRIPTION:
Patients scheduled for elective colonoscopy for screening are enrolled. On the day of the procedure, demographic data are collected and all patients are asked to complete the Spielberger State-trait Anxiety Inventory (STAI-I and STAI-II) in an isolated, calm room before being transferred to the procedure room.

All patients are monitored with electrocardiogram, pulse oximetry, noninvasive blood pressure and bispectral index measurement at 5-min intervals.

Oxygen is administered at 4 L/min via a face mask, Propofol 2% infusion is started via an effect-site target controlled infusion system (Marsh model).

Once the patient reaches the desired level of sedation as determined by BIS value of 60, the procedure is started.

This monitorization and sedation protocol is the routine management of outpatient colonoscopies and gastroscopies in our institution.

For this study the patients' anxiety levels are evaluated with the STAI score. This is not an intervention but an evaluation of the patients. Drug dosing or sedation management are not adjusted according to the anxiety scores but are calculated with the patients' weight.

During the procedure:

* hemodynamic parameters
* the total propofol dosage
* the number of TCI interventions
* complications (respiratory depression, need for ventilation, nausea, vomiting, laryngospasm, and agitation)
* the procedure duration
* surgeon satisfaction with sedation instrument scores are recorded.

These collected data are studies to determine a correlation between the propofol dose and the pre-procedural anxiety of the patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology Physiologic assessment score I-II patients
* 18-65 years old
* planned elective colonoscopy under sedation

Exclusion Criteria:

* the use of anxiolytic medications
* history of colonic resection or any intraabdominal surgery
* predicted allergy to propofol
* patients refusing sedation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 75 healthy patients undergoing elective colonoscopies as a screening test.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of pre-procedural anxiety level on the dose of propofol needed for sedation during the procedure. | The anxiety of all patients is evaluated at the day of the procedure. The procedure is then performed under sedation. Once the procedure is ended and all patients are fully awake, study data are collected and patients are discharged home.
  The sedation protocol applied in this study is our routin approach for all outpatient colonoscopies and endoscopies. All patients are informed about the procedures and monitorized (EKG, spO2, Bispectral index, blood pressure). After that, the sedation protocol is started and once the appropriate BIS value is reached the procedure is started. For this study all patients were asked to complete the STAI scores to evaluate the pre-procedural anxiety. This is not an intervention but an evaluation of the patients' anxiety. The primary outcome measure is to evaluate the dose of propofol used in each patient and to find out if there is a correlation between the pre-procedural anxiety and the dose of propofol.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Ceyda MECO, MD, DESA, Principal Investigator — Ankara University Faculty of Medicine; Mehmet Ayhan Kuzu, Prof, Study Director — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ibni Sina Hospital colonoscopy lab, Ankara, Turkey (Türkiye)